CLINICAL TRIAL: NCT05553873
Title: Evaluation of Inflammatory Markers in ph Negative Myeloproliferative Neoplasms: Impact on Outcome and Response to Therapy. Multicenter Retro-prospective Observational Study. The INFLA-ME (INFLAmmation in Myeloproliferative Disease) Study.
Status: Recruiting | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: INFLA-ME
Record Dates: First submitted 2022-09-21; First posted 2022-09-23 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Myeloproliferative Disease; Inflammatory Markers
MeSH Terms: conditions — Myeloproliferative Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to observe inflammatory biomarkers and their trend over the history of the disease in patients suffering from MPN Ph negative; it also wants to identify any correlations between the aforementioned biomarkers and disease outcomes, considering first of all the occurrence of thrombo-haemorrhagic events and the evolution in the accelerated / blast phase of the disease, shedding light on new tools that can potentially guarantee a prompt and better risk stratification

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of diagnosis of MPN Ph negative
* Diagnosis of PV, ET, PMF or post PV and post ET MF, according to current WHO or IWG-MRT criteria (diagnosis since 2000)
* Obtaining informed consent

Exclusion Criteria:

* Life expectancy of less than 6 months
* Accelerated phase myelofibrosis or MPN with signs of leukemic evolution

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults diagnosed with PV, ET, PMF or post PV and post ET MF, according to current WHO or IWG-MRT criteria (diagnosis since 2000)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-09-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
CBC with leukocyte formula and calculation of the NLR and PLR ratio | 60 months
Occurrence of arterial and venous thrombotic events | 60 months
  type of event, time to event after diagnosis, during illness

SECONDARY OUTCOMES:
Measurement of new and conventional inflammatory biomarkers | 60 months
  at the occurrence of the transformation in the overt phase from pre-fibrotic phase in the setting of myelofibrosis or at the occurrence of the evolution of the MPN Ph negative disease in an accelerated and / or leukemic phase or after 6 months from the introduction of conventional cytoreduction or target-therapy ( JAk2 inhibitors) or 6 months after the introduction of inflammatory drugs (iron chelators)
Time to thrombo-haemorrhagic events | 60 months
Time to death and been alive at the end of the study | 60 months
Time to evolution of the PH negative MPN disease into the fibrotic, accelerated or leukemic phase | 60 months

CONTACTS AND LOCATIONS:
Locations (11):
- Italy (11):
  - Azienda Ospedaliera Universitaria Consorziale Policlinico, Bari
  - Policlinico Sant'Orsola Malpighi, Bologna
  - ASST Spedali Civili di Brescia, Brescia
  - Policlinico Vittorio Emanuele, Catania
  - Ospedale Universitario Federico II, Napoli
  - Policlinico Umberto I, Università La Sapienza, Roma
  - Azienda Ospedaliera Universitaria Città della Salute e delle Scienza, Torino
  - Ospedale San Luigi di Orbassano - Ospedale Mauriziano, Torino
  - Azienda Ospedaliera Universitaria Friuli Centrale, Udine
  - Azienda Ospedaliera Universitaria Integrata, Verona
  - Ospedale Belcolle, Viterbo